CLINICAL TRIAL: NCT04032873
Title: Influence of Cost Information on Cast vs. Splint Decision-Making After Pediatric Buckle Fractures: A Randomized Controlled Trial
Brief Title: Distal Radius Buckle Fracture RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-013965
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Distal Radius Fracture
Keywords: Distal Radius Fracture; Cost; Buckle Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Provider Cost (Other): The subject will be given information about the cost of casting and splinting for treatment of the buckle fracture by the orthopaedic surgeon before the decision for immobilization has been made.
  Interventions: Other: Monetary Cost of Immobilization Treatments; Other: Physician; Other: Before Initial Treatment Decision
- Research Team Cost (Other): The subject will be given information about the cost of casting and splinting for treatment of the buckle fracture by a member of the study team after the decision for immobilization has been made.
  Interventions: Other: Monetary Cost of Immobilization Treatments; Other: Study Team; Other: After Initial Treatment Decision

INTERVENTIONS:
Other: Monetary Cost of Immobilization Treatments — Information regarding the monetary cost of casting and splinting patient's buckle fracture to be presented to adult subject/payer.
  Other Names: Cost Information
Other: Physician — The monetary cost information is relayed by the patient's physician
  Arms: Provider Cost
Other: Study Team — The monetary cost information is relayed by a member of the study team
  Arms: Research Team Cost
Other: Before Initial Treatment Decision — Monetary cost information is relayed during the initial consult, before the treatment decision is made.
  Other Names: Initial Consult
  Arms: Provider Cost
Other: After Initial Treatment Decision — Monetary cost information is relayed after the initial consult with the treating physician, after the treatment decision is made.
  Other Names: Post-Consult
  Arms: Research Team Cost

SUMMARY:
This study evaluates the influence of cost information on decision-making for immobilization for treatment of distal radial buckle fractures. Half of the participants will receive cost information from an orthopaedic surgeon prior to making their decision for treatment, while the other half will receive cost information from another member of the study team after they had made their decision treatment.

DETAILED DESCRIPTION:
Research has shown equipoise in treatment outcomes after casting and splinting for pediatric buckle fractures. Despite the similarly favorable treatment outcomes associated with both casting and splinting these fractures, there is wide disparities in cost between the two types of immobilization. However, cost information is not routinely presented to families during the discussion of immobilization types.

The primary objective of this study is to determine if cost information influences family decision-making about immobilization type after pediatric buckle fractures. A secondary objective is to determine if the timing of and person disseminating the cost information changes the influence it has on families' decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 4 to 14 years with a buckle fracture for which they will be treated with a cast or a splint.
* Parental/guardian permission (informed consent) and, if appropriate, child assent.
* Parent of a child ages 4 to 14 years with a buckle fracture that requires treatment with either a cast or a splint.
* Parental/guardian permission (informed consent).

Exclusion Criteria:

* Non-English speaking subjects.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Monetary Cost of Immobilization's Influence on Treatment Decisions | 1 to 5 minutes
  The outcome measure will evaluate whether monetary cost influenced payers' decisions to choose one immobilization treatment over the other (splinting vs. casting).

SECONDARY OUTCOMES:
Timing/Person Effect on Decision-Making | 1 to 5 minutes
  A secondary objective is to determine if the timing of and person disseminating the cost information changes the influence it has on families' decision-making

CONTACTS AND LOCATIONS:
Overall Officials: John Todd R Lawrence, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with researchers outside of the research team for this clinical trial.